CLINICAL TRIAL: NCT04384003
Title: Integrated Proximal and Distal Joint Exercise Therapy Interventions on the Performance and Injury Prevention in Competitive Sports: Effects of Motor Control and Tissue Biomechanics
Brief Title: Integrated Exercise Therapy Interventions on the Performance and Injury Prevention in Competitive Sports
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P00000801
Record Dates: First submitted 2020-04-21; First posted 2020-05-12 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Strain of Fascia of Intrinsic Muscle of Foot (Disorder); Elastography; Muscle Weakness
Keywords: Foot core system; Muscle stiffness; Motor control; Shear wave ultrasound elastography; Electromyography
MeSH Terms: conditions — Muscle Weakness | interventions — Physical Examination

STUDY DESIGN:
Who Masked: Participant
Masking Description: a single-blinded randomized controlled trial will be conducted, in which patients will be randomized into groups by sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Shear Wave Ultrasound Elastography (Active Comparator): Shear Wave Ultrasound Elastography (SWUE, AplioTM 300 Platinum, Toshiba Medical System Corp, Japan, 6I) to examine the morphology and mechanical properties (μ = ρVs2, μ is the shear modulus of the tissue, ρ is the density of muscle (1000 kg m-3), Young's modulus )
  Interventions: Device: Shear Wave Ultrasound Elastography; Device: The 3-D Motion Analysis; Device: Electromyographic; Diagnostic Test: Foot intrinsic muscle assessment and training device
- The 3-D Motion Analysis (Active Comparator): An optoelectronic-based 3D motion analysis system, including cameras, force plates, and an EMG system will be used in this study. A lower limb model (pelvis included) will be established through commercial motion analysis software (VICON Corp, UK). We will use this model to measure joint kinematics, joint kinetics, and ground reaction forces during functional activities, such as level walking.
  Interventions: Device: Shear Wave Ultrasound Elastography; Device: The 3-D Motion Analysis; Device: Electromyographic; Diagnostic Test: Foot intrinsic muscle assessment and training device
- EMG acquisition system (Active Comparator): Electromyographic signals measures will be focused on the Abductor Hallucis (AbdH), Peroneus Longus (PL) and Previous Brevis (PB), Gluteus Medius (Glut Med), and Gluteus Maximus (Glut Max). In order to reduce the cross-talk of other muscles in the foot, a miniature wireless surface EMG sensor (TrignoTM Mini Sensor, Delsys Inc. USA) will be used after confirmation of our previous research results.
  Interventions: Device: Shear Wave Ultrasound Elastography; Device: The 3-D Motion Analysis; Device: Electromyographic; Diagnostic Test: Foot intrinsic muscle assessment and training device
- Foot intrinsic muscle assessment and training device (Active Comparator): Schematic diagram of the novel modified foot intrinsic muscle (FIM) assessment and training device, which consists of one controller unit (signal generators, amplifier and A/D converter; signal generators provide noise-enhanced vibration to facilitate the muscle activation), 2 voice coil motor & server, 2 optical rulers, 2 rail scale, and 7 load cells.
  The main concept for this design is to provide the quantitative assessment of the foot intrinsic muscles and facilitation of intrinsic muscles of the fool during functional sporting activities such single-leg-standing and kicking.
  Interventions: Device: Shear Wave Ultrasound Elastography; Device: The 3-D Motion Analysis; Device: Electromyographic; Diagnostic Test: Foot intrinsic muscle assessment and training device

INTERVENTIONS:
Device: Shear Wave Ultrasound Elastography — Scanned protocols of sonographic imaging will be used in this study to measure extrinsic (FDL, FHL and PER) and intrinsic (AbdH, FDB and FHB) muscle CSA and thickness, and plantar fascia thickness (at heel, mid and forefoot sites).
  The muscle stiffness will be calculated from the program provided by the US machine as shown real time elastography (RTE, unit: KPa).
  Other Names: AplioTM 300 Platinum
Device: The 3-D Motion Analysis — The 3-D Motion Analysis, Forceplates and EMG acquisition system and full body kinematic model (Bonita, VICON Corp, UK) in the Biomechanics and Motor Control Laboratory (BMCL).
  Other Names: Bonita, VICON Corp, UK,
Device: Electromyographic — Electromyographic activity (EMG) of AbdH, TA, PL, SO, gluteus medius (Glut Med) and gluteus maximus (Glut Max) will be recorded bilaterally using pairs of surface electrodes. Motor coordination of these muscles will be evaluated through assessment of temporal and spatial parameters of EMG during functional tasks such as kicking in one leg standing. The primary outcome measure will be percentage of EMG relative to maximal voluntary contraction (MVC) on the same side. In order to remove the potential for investigator bias, all data will be presented individually without identification of the muscle, order of trials or whether the trials precede or follow the intervention.
  Other Names: TrignoTM, Delsys Corp. USA
Diagnostic Test: Foot intrinsic muscle assessment and training device — The main concept for this design is to provide the quantitative assessment of the foot intrinsic muscles and facilitation of intrinsic muscles of the fool during functional sporting activities such single-leg-standing.
  Other Names: Schematic diagram of the novel modified foot intrinsic muscle (FIM) assessment and training device

SUMMARY:
Football is an increasingly popular exercise and common practice among adolescent and elite athletes. However, these athletes tend to have injuries involving the lower extremity and foot. Recent literature has proposed a promising concept of core stability on the arch of the foot and proximal hip control exercise for a knee injury. They have highlighted that foot core training begins with targeting the plantar intrinsic muscles through exercise intervention, which may enhance the capacity and control of the foot core system. Moreover, it is hypothesized that the 'complexity algorithm' of exercise intervention for proximal hip control may provide more sufficient effects on musculoskeletal pain in the lower extremity. However, some conflicting issues such as assessment and training of foot intrinsic muscle in functional positions still largely lack devices and research to elucidate the underlying mechanism of its development and integrated exercise interventions proximally and distally on these athletes.

Firstly, the investigators aim to design and develop of novel intrinsic foot muscle assessment and training device for sporting tasks and to examine the feasibility and reliability of muscle stiffness in foot and hip joints before and after exercise intervention using shear wave ultrasound elastography (SWUE) in athletes without and with foot and ankle overuse injuries; second, investigators will investigate whether immediate and persistent alteration after the integrated therapeutic exercise on motor control and muscle stiffness.

DETAILED DESCRIPTION:
The foot often plays a crucial role in sensorimotor control and movement performance in standing, walking, and running. Anatomically, the intrinsic foot muscles (IFM) are the primary local stabilizer to provide static and dynamic stability in the foot, which are part of the active and neural subsystems to constitute the foot core system. The intrinsic foot muscles (IFMs) may play a key role in supporting foot arches (e.g. the medial longitudinal arch, MLA), providing flexibility, stability, shock absorption to the foot, and partially controlling foot pronation. Due to the difficulties in teaching and learning the plantar intrinsic foot muscle (IFM) exercise, the accuracy and follow-up after learning this exercise could be questioned following this exercise program; Physiologically, the effects of exercise intervention may be achieved following more than 4-week intensive exercise intervention at least. How to learn and activating this kind of exercise efficiently and effectively is key for employing this exercise in young athletes with and without flexible flat feet.

This project consists of two main parts - first, we aim to design and develop of novel intrinsic foot muscle strengthening device using 3-D printing techniques and to examine the feasibility and reliability of the morphology and neuromotor control features in intrinsic and extrinsic foot muscles before and after exercise intervention using Transcranial Magnetic Stimulation (TMS) and sonographic imaging in football /basketball athletes with without flexible flat feet (FFF); second, we will investigate whether immediate and persistent alterations in the morphology and motor control of IFMs and dynamic postural control after this therapeutic exercise with novel 3-D printing foot core exerciser. More importantly, we also elucidate important clinical evidence-based information on long-term novel therapeutic exercise intervention for coaches, clinicians, and health policymakers.

ELIGIBILITY:
Inclusion Criteria:

Athletes with plantar heel pain:

1. Diagnosis of painful heel syndrome by clinical examination, with the following positive clinical signs:

   1. Pain in the morning or after sitting a long time
   2. Local pain where the fascia attaches to the heel
   3. Increasing pain with extended walking or standing for more than 15 minutes
2. Was associated with inflammatory symptoms (pain, swelling, etc.)
3. Pain in the area of the insertion of the plantar aponeurosis on the medial tubercle of the calcaneus.
4. Not perform ankle stretching exercises as treatment of the plantar fasciitis.

Healthy individuals:

1. A neutral foot alignment: determined by measurement of the resting calcaneal stance position (RCSP: between 2°of inversion and 2°of eversion) and scores on the navicular drop (ND: between 5 and 9 mm) test.
2. Foot Posture Index Score is between 0 and 5 .
3. No pain in the lower limbs
4. No history of lower limb injury or surgery that has affected function or caused the Individual to seek previous medical or therapeutic intervention.

Exclusion Criteria:

1. Traumatic injury to lower limbs which impacted joint integrity and function (i.e., fractures) resulting in at least 1 interrupted day of desired physical activity
2. History of spinal, pelvic or lower limb surgery
3. Major neurological, cardiorespiratory or circulatory disorders
4. Past history of traumatic head injury with or without loss of consciousness
5. Have been taking non-steroidal anti-inflammatory or corticosteroid medication in the past month
6. Recent intervention/management within the last 6 months

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area (CSA) | 6 months
  Parameters of morphology (CSA) of intrinsic and extrinsic foot and selected hip muscles. The unit is cm².
Cross-sectional area (CSA) | 12 months
  Parameters of morphology (CSA) of intrinsic and extrinsic foot and selected hip muscles. The unit is cm².
Thickness | 6 months
  Parameters of morphology (thickness) of intrinsic and extrinsic foot and selected hip muscles. The unit is cm.
Thickness | 12 months
  Parameters of morphology (thickness) of intrinsic and extrinsic foot and selected hip muscles. The unit is cm.
Stiffness (RTE) | 6 months
  Parameters of morphology Stiffness (RTE) of intrinsic and extrinsic foot and selected hip muscles. The unit is kPa.
Stiffness (RTE) | 12 months
  Parameters of morphology Stiffness (RTE) of intrinsic and extrinsic foot and selected hip muscles. The unit is kPa.
Joint kinematics and joint kinetics in the hip, knee and ankle joints will be calculated with the data | 12 months
  Biomechanical data (i.e. joint kinematics such as joint angle and joint kinetics such as joint moments in the lower limb), center of pressure (CoP, i.e. the trajectory curve) and center of mass (CoM, i.e. the trajectory curve ) and electromyographic data (unit, percentage of maximal voluntary isometric contraction, MVIC) will be analyzed, respectively. Joint kinematics and joint kinetics in the hip, knee and ankle joints will be calculated with the data integrated from motion capture system (Nexus 2.0, Bodybuilder 3.6.4, Vicon Corp. UK ) and forceplates (Kistler, 9286B, Switzerland).
Joint kinematics and joint kinetics in the hip, knee and ankle joints will be calculated with the data | 6 months
  Biomechanical data (i.e. joint kinematics such as joint angle and joint kinetics such as joint moments in the lower limb), center of pressure (CoP, i.e. the trajectory curve) and center of mass (CoM, i.e. the trajectory curve ) and electromyographic data (unit, percentage of maximal voluntary isometric contraction, MVIC) will be analyzed, respectively. Joint kinematics and joint kinetics in the hip, knee and ankle joints will be calculated with the data integrated from motion capture system (Nexus 2.0, Bodybuilder 3.6.4, Vicon Corp. UK ) and forceplates (Kistler, 9286B, Switzerland).
Electromyographic(EMG) | 6 months
  Electromyographic variables (IEMG) between individuals with and without plantar heel pain (PHP) will be compared using a repeated-measures analysis of variance.measures analysis of variance
Electromyographic(EMG) | 12 months
  Electromyographic variables (IEMG) between individuals with and without plantar heel pain (PHP) will be compared using a repeated-measures analysis of variance.measures analysis of variance

CONTACTS AND LOCATIONS:
Overall Officials: Chich-Haung R. Yang, PhD, Principal Investigator — College of Medicine, Tzu Chi University
Locations (1):
- BuddhistTCGH, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No